CLINICAL TRIAL: NCT02341313
Title: Feasibility of the Use of Point of Care Technology to Measure Ketone and Lactate Levels in the Newborn at Risk From Hypoglycaemia Due to Impaired Perinatal Counter Regulation
Brief Title: Point of Care Ketone Measurement in the Newborn
Acronym: POCKET
Status: Completed | Type: Observational
Sponsor: Kathryn Beardsall (Other)
Responsible Party: Sponsor-Investigator, Kathryn Beardsall, University Lecturer Consultant Neonatologist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 13/EE/0443
Record Dates: First submitted 2014-03-16; First posted 2015-01-19 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Hypoglycaemia
Keywords: Hypoglycaemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newborns at risk of hypoglycaemia: Measurement of ketones

SUMMARY:
Low blood sugar levels are common in babies after birth. This may be normal as babies can use other sources of energy. However if a baby does not produce these fuels the brain can be starved of energy and be damaged. Measurement of these fuels is not done as part of clinical practice in the newborn. The investigators aim to see whether at the same time as taking the blood sugar level from a heel prick these fuels can be measured in a small drop of blood. At the same time as blood needs to be taken for clinical reasons the study team will to take a drop of blood from 50 babies to see how good the point of care (POC) meters are compared to the laboratory at measuring these fuels. If accurate these POC meters could identifying those at risk from brain damage as well as prevent separation of mothers and babies who are establishing breast feeding.

ELIGIBILITY:
Inclusion Criteria:

* Infants having blood samples taken for clinical management of glucose control

Exclusion Criteria:

-

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants at risk of hypoglycaemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Measure of ketone levels between Point of care and laboratory assessment | Neonatal period up to 28 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Beardsall, MRCP, Principal Investigator — Cambridge University
Locations (1):
- addenbrookes Hospital, Cambridge, United Kingdom